CLINICAL TRIAL: NCT03051503
Title: Efficacy of Transdermal Fentanyl Patches in Relief of Acute Postoperative Pain After Mastectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Dr.mohamad farouk mohamad, lecturer of anesthesia and pain relief, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 228
Record Dates: First submitted 2017-02-03; First posted 2017-02-13 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The Transdermal Therapeutic System-Fentanyl (TTS-F) group (Active Comparator): (TTS-F) group (n=30) 50ug/h patch, placed 12 hs preoperatively.
  Interventions: Drug: The Transdermal Therapeutic System-Fentanyl (TTS-F)
- Intravenous patient-controlled analgesia (PCA) morphine (Placebo Comparator): IV (PCA) morphine for pain in the postoperative period.
  Interventions: Device: Intravenous patient-controlled analgesia (PCA) morphine

INTERVENTIONS:
Drug: The Transdermal Therapeutic System-Fentanyl (TTS-F) — (TTS-F) group (n=30) 50ug/h patch, placed 12 hours preoperatively
  Other Names: Fentanyl patch
  Arms: The Transdermal Therapeutic System-Fentanyl (TTS-F) group
Device: Intravenous patient-controlled analgesia (PCA) morphine — IV PCA morphine for pain in the postoperative period.
  Other Names: IV PCA morphine
  Arms: Intravenous patient-controlled analgesia (PCA) morphine

SUMMARY:
to determine the safety, efficacy and tolerability of transdermal fentanyl in patients undergoing mastectomy, as well as the postoperative consumption of analgesic.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II patients
* aged 30-60 years
* body weight ranged between 65-10kg

Exclusion Criteria:

* Patients with history of allergy to morphine
* chronic intake of analgesics or non-steroidal anti-inflammatory drug 24 h prior to surgery,
* there was a history of a psychiatric disorder patients weight was less then 50kg.
* impaired kidney function.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Total dose of morphine consumption in the first 48 hours postoperative | 48 hours
  Total dose of I.V. PCA morphine consumption in the first 48 hours postoperative
Visual Analogue Scale | 48 hours
  Pain measurement scale

SECONDARY OUTCOMES:
Level of stress hormones | 48 hours
  Cortisol levels
Side effects related to the opioids | 48 hours
  Nausea and vomiting; Itching; Respiratory depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Othman, MD, Study Director — Cancer Institute, Anesthesia, Intensive Care, and Pain Management, South Egypt Cancer Institute, Assiut University, Assiut, Egypt
Locations (1):
- South Egypt Cancer Institute, Assiut University, Assiut, Egypt., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes